CLINICAL TRIAL: NCT01862081
Title: A Dose-escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of GDC-0032 in Combination With Docetaxel or With Paclitaxel in Patients With HER2-negative Locally Recurrent or Metastatic Breast Cancer or Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO27802; 2013-003543-28 (EudraCT Number)
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer, Non-small Lung Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm A: GDC-0032 + Docetaxel (Experimental): Participants will receive GDC-0032 once daily for 21 consecutive days (beginning from Day 1) in each 21-day cycle along with Docetaxel on Day 1 of each 21-day cycle.
  Interventions: Drug: Docetaxel; Drug: GDC-0032
- Arm B: GDC-0032 + Paclitaxel (Experimental): Participants will receive GDC-0032 once daily for 28 consecutive days (beginning from Day 1) in each 28-day cycle along with Paclitaxel on Days 1, 8, 15 and 22 of each 28-day cycle.
  Interventions: Drug: GDC-0032; Drug: Paclitaxel
- Arm C: GDC-0032 + Docetaxel (Experimental): Participants will receive GDC-0032 once daily on Day 1 and Days 8-14 of each 21-day cycle along with Docetaxel on Day 1 of each 21-day cycle.
  Interventions: Drug: Docetaxel; Drug: GDC-0032
- Arm D: GDC-0032 + Docetaxel (Experimental): Participants will receive GDC-0032 once daily on Days 2-14 of each 21-day cycle along with Docetaxel on Day 1 of each 21-day cycle.
  Interventions: Drug: Docetaxel; Drug: GDC-0032
- Arm E: GDC-0032 + Docetaxel (Experimental): Participants will receive GDC-0032 once daily on Days 1-14 of each 21-day cycle along with Docetaxel on Day 1 of each 21-day cycle.
  Interventions: Drug: Docetaxel; Drug: GDC-0032
- Arm F: GDC-0032 + Paclitaxel (Experimental): Participants will receive GDC-0032 once daily on a 5-days on, 2-days off schedule in each 28-day cycle along with Paclitaxel on Days 1, 8, 5 and 22 of each 28-day cycle.
  Interventions: Drug: GDC-0032; Drug: Paclitaxel
- Arm G: GDC-0032 + Paclitaxel (Experimental): Participants will receive GDC-0032 once daily on a 3-days on, 4-days off schedule in each 28-day cycle along with Paclitaxel on Days 1, 8, 5 and 22 of each 28-day cycle.
  Interventions: Drug: GDC-0032; Drug: Paclitaxel

INTERVENTIONS:
Drug: Docetaxel — Participants will receive docetaxel 75 milligrams per meter-squared (mg/m^2) intravenous (IV) dose on Day 1 of each 21-day cycle.
  Arms: Arm A: GDC-0032 + Docetaxel; Arm C: GDC-0032 + Docetaxel; Arm D: GDC-0032 + Docetaxel; Arm E: GDC-0032 + Docetaxel
Drug: GDC-0032 — Participants will receive escalated dose of GDC-0032. The initial dose will be 3 mg capsules or 2 mg tablets.
Drug: Paclitaxel — Participants will receive paclitaxel 80 mg/m^2 IV dose on Day 1, 8, 15 and 22 of each 28-day cycle.
  Arms: Arm B: GDC-0032 + Paclitaxel; Arm F: GDC-0032 + Paclitaxel; Arm G: GDC-0032 + Paclitaxel

SUMMARY:
This is an open-label, multicenter, dose-escalation study designed to assess the safety, tolerability, and pharmacokinetics of oral GDC-0032 administered in combination with either docetaxel or with paclitaxel. Patients treated with the GDC-0032 and docetaxel have HER2-negative locally recurrent or metastatic breast cancer or non-small cell lung cancer (NSCLC). Patients treated with the GDC-0032 and paclitaxel combination have human epidermal growth factor receptor 2 (HER2)-negative locally recurrent or metastatic breast cancer. There are two potential stages within each arm of this study: a dose-escalation stage (Stage 1) and a dose-expansion stage (Stage 2). Once the maximum tolerated dose of GDC-0032 in a given arm has been established from dose escalation, additional patients with each combination will be enrolled in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* For paclitaxel combination arms: histologically or cytologically documented adenocarcinoma of the breast with locally recurrent or metastatic disease
* For docetaxel combination arms: histologically or cytologically documented adenocarcinoma of the breast with locally recurrent or metastatic disease or histologically documented advanced (Stage IV) or recurrent NSCLC
* For participants with breast cancer: HER2-negative disease as defined by local clinical guidelines
* Participants with NSCLC to be treated with docetaxel need to have received at least one prior anti-cancer treatment regimen in an advanced setting and to have docetaxel be considered appropriate treatment
* Evaluable or measurable disease per response evaluation criteria in solid tumors (RECIST) v.1.1
* Life expectancy >=12 weeks
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1 at screening
* Adequate hematologic and end organ function
* Use of highly effective form of contraception

Exclusion Criteria:

* Prior anti-cancer therapy
* Prior treatment with phosphoinositide 3-kinase (PI3K) inhibitor
* Known significant hypersensitivity to any components of study treatment
* Grade >=2 peripheral neuropathy
* Type 1 or Type 2 diabetes
* Grade >=2 hypercholesterolemia or hypertriglyceridemia
* Congenital long QT syndrome
* Active congestive heart failure or ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07-16 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | Approximately 3 years
Safety: Incidence of dose limiting toxicities | Up to 28 days

SECONDARY OUTCOMES:
Area under the curve from time 0 to the last measurable concentration (AUC0-last) | Up to 28 days
Time to maximum observed plasma concentration (Tmax) | Up to 28 days
Maximum observed plasma concentration (Cmax) | Up to 28 days
Minimum observed plasma concentration (Cmin) | Up to 28 days
Objective response according to RECIST v1.1 | Approximately 3 years
Duration of response according to RECIST v1.1 | Approximately 3 years
Progression-free survival (PFS) according to RECIST v1.1 | Approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (14):
- United States (10):
  - Florida Cancer Specialists - Tampa (Dr. MLK Blvd), Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, P.A; Baylor Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, P.A. - Fort Worth, Fort Worth, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
- UZ Leuven; Maag, -darm en leverziekten/endoscopie - Endoscopy, Leuven, Belgium
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinico Universitario de Valencia, Valencia